CLINICAL TRIAL: NCT04590157
Title: Neuromodulation Effect of Laser Acupuncture on Female Stress Urinary Incontinence: A Randomized Controlled Trial
Brief Title: Neuromodulation Effect of Laser Acupuncture on Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lama Saad El-Din Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Lama Saad El-Din Mahmoud, Lecturer of physical therapy, Department of Neuromuscular disorders and its surgery, faculty of physical therapy, october 6 univerisity, October 6 University
Organization: October 6 University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T. REC/012/002930
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Stress Urinary Incontinence
Keywords: Neuromodulation; laser acupuncture; neurogenic acupoints; female stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: the control group received pelvic floor muscle training ,and the study group received the same program in addition to laser acupuncture on neurogenic acupoints
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): received pelvic floor muscle training in addition to laser acupuncture on neurogenic acupoints
  Interventions: Device: Low Level Laser Therapy; Other: Pelvic floor muscle training
- control group (Experimental): received pelvic floor muscle training
  Interventions: Other: Pelvic floor muscle training

INTERVENTIONS:
Device: Low Level Laser Therapy — Laser Acupuncture application on Neurogenic Acupoints: the treatment based upon the use of low power laser light to stimulate acupuncture points
  Arms: study group
Other: Pelvic floor muscle training — exercise prodram as follow: from supine lying position with legs slightly apart the patient asked to contract the pelvic muscles as hard as possible and hold for 10 seconds

SUMMARY:
background:Stress urinary incontinence (SUI) is the most common type of urinary incontinence in women, as it involves involuntary leakage of urine , the current study was To determine the neuromodulation effect of Laser Therapy on Neurogenic Acupoints in female with stress urinary incontinence (SUI).

DETAILED DESCRIPTION:
Thirty women with SUI were randomly divided into two equal groups; the control group received pelvic floor muscle training , while the study group received the same pelvic floor muscle training in addition to laser acupuncture on neurogenic acupoints . The outcome measures were pelvic floor muscle strength (PFMS) , SUI severity assessed by Severity Index (SI) , and Incontinence Questionnaire-Short Form (ICIQ-SF). The outcome measures were assessed pre- and post-rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* age ranged from 30 to 45 years old
* body mass index (BMI) was less than 30 kg/m2,
* all women were non-smokers and they had a sedentary life style

Exclusion Criteria:

* The participants were excluded if they had other types of urinary incontinence (urge or mixed)
* urinary tract infection
* pelvic organ prolapse
* diabetes mellitus
* respiratory diseases, chronic cough and constipation

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor muscle strength (PFMS) | 6 weeks
  The pelvic floor muscle strength of all women in both groups was assessed pre- and post-rehabilitation program, using XFT-0010 Pelvic Muscle Trainer device
Stress urinary incontinence (SUI) severity | 6 weeks
  The incontinence severity index (ISI) consists of two questions, regarding frequency and amount of leakage. It categorizes urinary incontinence (UI) into slight, moderate, severe, and very severe.
International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF). | 6 weeks
  it is a validated subjective measure used to assess the Stress urinary incontinence and its impact on quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A Osman, PHD, Principal Investigator — lecturer, department of physical therapy for Women's Health faculty of physical therapy ,Cairo university,Egypt; Khadiga S Abdulaziz, Study Director — professor,department of physical therapy for Women's Health faculty of physical therapy ,Cairo university,egypt; Doha R Ahmed, Bachelor, Principal Investigator — Department of Physiotherapy, Ahmed Maher Teaching Hospital, Cairo, Egypt; Emad E Atiya, PHD, Principal Investigator — Professor, Department of Urology, Ahmed Maher Teaching Hospital, Cairo, Egypt; Lama S Mahmoud, PHD, Principal Investigator — Lecturer, Department of Physical Therapy For Neuromuscular Disorders and its surgery, Faculty of Physical Therapy, October 6 University, Egypt
Locations (1):
- October 6 University, Giza, El-Sheikh Zayed City Giza 1133 Egypt, Egypt